CLINICAL TRIAL: NCT02469467
Title: A Dose Escalation Study of VS-505 to Evaluate the Tolerability, Safety and Efficacy in End Stage Renal Disease Patients Undergoing Hemodialysis
Brief Title: A Dose Escalation Study of VS-505 in End Stage Renal Disease Patients Undergoing Hemodialysis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KDL Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VDKDL001
Record Dates: First submitted 2015-06-01; First posted 2015-06-11 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: End Stage Renal Disease; Hyperphosphatemia
Keywords: phosphate binder; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VS-505 (Experimental): 750 mg capsule
  Interventions: Dietary Supplement: VS-505

INTERVENTIONS:
Dietary Supplement: VS-505 — VS-505 is orally administered with meal for 8 weeks

SUMMARY:
The purpose is to evaluate the tolerability, safety and efficacy of VS-505 when given with meal for 8 weeks to hemodialysis patients with hyperphosphatemia

DETAILED DESCRIPTION:
This study consists of 4 period; 1) screening period: up to 30 days, 2) first washout period: 2 weeks (remove existing phosphate binder effect), 3) treatment period: 8 weeks, and 4) second washout period: 2 weeks (remove VS-505 effect). VS-505 is orally administered with meal for 8 weeks. The starting dose of VS-505 is 1.50 g/day and the dose will be elevated step wise from 1.50 g to 2.25 g, 4.50 g and 6.75 g per day based on the safety assessment and plasma Pi level every 2 weeks during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given
* Able to comply with the study procedures and medications
* On a stable hemodialysis (HD) regimen (3 times per week) including hemodialysis and hemodiafiltration for ≥12 weeks at screening and during the study period
* No change in prescribed dose or frequency of any of the following medications within 4 weeks prior to screening

  1. Injectable iron agents
  2. Oral or injectable active vitamin D3
  3. Oral nutritional vitamin D
  4. Calcimimetics
  5. Calcium supplements
  6. Anti-osteoporotic medication including bisphosphonates
  7. Calcitonins
* Must be willing to avoid intentional changes in diet throughout the study
* Women of child-bearing potential or non-sterile male subjects and those who are sexually active with a non-sterile female partner must agree to use highly effective contraception
* Plasma Pi level >1.94 mmol/L (6.0 mg/dL) to <3.23 mmol/L (10.0 mg/dL) after 2 weeks washout will qualify patients to enter the treatment period

Exclusion Criteria:

* Blood purification therapy other than HD (hemodialysis and hemodiafiltration)
* The plasma Pi level is >2.26 mmol/L (7.0 mg/dL) within the latest three tests prior to screening.
* Variation of the plasma Pi is over 0.65 mmol/L (2.0 mg/dL) within the latest three tests prior to screening.
* Pre-emptive or scheduled renal transplant
* History of hemochromatosis or ferritin ≥1000 mcg/L
* Oral iron agents including prescribed and over-the-counter drugs at screening.
* Current clinically significant gastrointestinal (GI) disorder, including GI bleeding, colitis, inflammatory bowel disease, irritable bowel syndrome, chronic constipation, new diagnosis of peptic or duodenal ulcer disease, within 4 weeks prior to screening
* History of gastrectomy or duodenectomy, or GI tract surgery within 12 weeks prior to screening
* Hypertension: Defined using pre-dialysis vital of diastolic blood pressure >110 mmHg or systolic blood pressure >180 mmHg
* Possible parathyroid intervention including surgical parathyroidectomy and percutaneous ethanol injection therapy during the study period
* Clinical evidence of active malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous carcinoma of the skin
* Severe cardiovascular disorders such as recent myocardial infarction; unstable angina; congested heart failure (NYHA class II or above) hospitalized within 24 weeks (6 months), valve stenosis, atrial fibrillation and arrhythmia
* History of event by cerebrovascular disease or cardiovascular disease within 24 weeks (6 months) prior to screening
* Active infection or current treatment with antibiotics within 2 weeks prior to screening
* History of HIV (ELISA and Western blot) test results
* Known active liver disease with aspartate aminotransferase or alanine aminotransferase levels greater than x3 the upper limit of normal
* Hepatitis B and/or hepatitis C treated with antiviral treatment within 4 weeks prior to screening
* History of allergy of VS-505 and its related components
* Receipt of any investigational drug within 4 weeks prior to screening
* Pregnant and breast-feeding women
* Other patients who in the opinion of the investigators are ineligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Inorganic phosphorus (Pi) change from baseline to end of treatment | 8 weeks

SECONDARY OUTCOMES:
Calcium (Ca) change from baseline to end of treatment | 8 weeks
Ca x Pi change from baseline to end of treatment | 8 weeks
intact parathyroid hormone change from baseline to end of treatment | 8 weeks
Rate of patients whose Pi reduction is 0.65 mmol/L (2.0 mg/dL) | 8 weeks
Rate of patients whose Pi reaches the goal between 1.13 mmol/L (3.5 mg/dL) and 1.94 mmol/L (6.0 mg/dL) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johan Rosman, MD, Ph.D, Principal Investigator — LCR Clinical Research
Locations (1):
- LCR Clinical Research, Perth, Western Australia, Australia